CLINICAL TRIAL: NCT06811662
Title: Outcomes of Complete Versus Partial Preservation of the Sub-valvular Apparatus in Cases of Mitral Valve Replacement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Mamdouh Hussein, dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: preservation of MV leaflts
Record Dates: First submitted 2024-12-07; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mitral Valve Replacement; Mitral Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- complete (preservation of both anterior and posterior leaflets) preservation of subvalvular apparatu (Active Comparator): complete (preservation of both anterior and posterior leaflets) preservation of subvalvular apparatus
  Interventions: Procedure: mitral valve replacement
- partial (preservation of posterior leaflet only) preservation of subvalvular apparatus (Active Comparator): partial (preservation of posterior leaflet only) preservation of subvalvular apparatus
  Interventions: Procedure: mitral valve replacement

INTERVENTIONS:
Procedure: mitral valve replacement — complete versus partial preservation of subvavular apparatus during mitral valve replacement

SUMMARY:
The purpose of this study is to evaluate the outcomes of complete (preservation of both anterior and posterior leaflets) versus partial (preservation of posterior leaflet only) preservation of subvalvular apparatus in cases of mitral valve replacement

DETAILED DESCRIPTION:
After mitral valve replacement (MVR), sudden increases in afterload and disruption of the annular-chordal-papillary-left-ventricular wall causes left ventricular (LV) dysfunction in the early postoperative period.

patients with LV dysfunction after MVR have a significantly lower 8-year survival rate compares with patients who did not have LV dysfunction Papillary muscles play an important role in the left ventricular contraction by drawing the mitral ring toward the apex, thereby causing shortening of the long axis and spherity of the chamber contribute for better ejection of blood.

preservation of papillary muscles and chordae tendineae in MVR reduces postoperative mortality, low cardiac output syndrome and improves haemodynamic function.

Partial preservation of the mitral apparatus through preservation of the posterior leaflet (MVR-P) has been proven to significantly reduce perioperative mortality.

The importance of complete preservation of the mitral apparatus remains controversial, but it is hypothesized that complete preservation with preservation of both the anterior and posterior leaflets may contribute to superior postoperative hemodynamic function as compared to partial preservation.

Due to the increased technical complexity of preserving both leaflets, concerns about longer bypass and cross-clamp times, the need to undersize prostheses, and the possibility of left ventricular outflow tract (LVOT) obstruction, the majority of cardiac surgeons currently prefer to preserve the posterior leaflet alone.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18 and 60 years
* Rheumatic mitral disease indicated for mitral valve replacement
* Concomitant other valve disease

Exclusion Criteria:

* - Patients who have undergone previous mitral valve surgery or other heart surgery.
* Patients with ischemic mitral disease.
* emergency operation.
* patients with significant comorbidities (severe pulmonary disease or end stage renal disease).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the outcomes of complete versus partial preservation of subvalvular apparatus in mitral valve replacement | anticepated 3 years
  To evaluate the outcomes of complete versus partial preservation of subvalvular apparatus in mitral valve replacement regarding:
  * Postoperative morbidity and mortality
  * LV function and the change of cardiac chamber dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Heart Hosiptal, Asyut, Egypt